CLINICAL TRIAL: NCT02346071
Title: Acceptance and Commitment Group Therapy for Adolescents With a Range of Functional Somatic Syndromes: Randomized Trial
Brief Title: Acceptance and Commitment Group Therapy for Adolescents With a Range of Functional Somatic Syndromes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Karolinska University Hospital (Other); National Research Centre for the Working Environment, Denmark (Other Government); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CURKHK1
Record Dates: First submitted 2014-12-02; First posted 2015-01-26 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Somatization Disorder; Somatoform Disorders
Keywords: Bodily distress syndrome; Medically unexplained symptoms; Functional somatic symptoms; Functional somatic syndromes; Treatment; Acceptance and Commitment Therapy
MeSH Terms: conditions — Somatoform Disorders; Medically Unexplained Symptoms | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced Usual Care (EUC) (Active Comparator): Clinical psychiatric and somatic assessment. Standard psychiatric consultation (SPC) given 2 weeks after randomization.
  Interventions: Other: Enhanced Usual Care (EUC)
- Acceptance and Commitment Therapy (ACT) (Experimental): Clinical psychiatric and somatic assessment. Standard psychiatric consultation (SPC) given 2 weeks after randomization. ACT-based group therapy.
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — All patients will have a thorough clinical psychiatric and somatic assessment in order to determine eligibility and a psychiatric consultation (SPC) of 1-1½ hrs. duration approx. 2 weeks after randomization.
  The ACT treatment is manualized and given in groups of 7-8 patients with 9 3-hour sessions (i.e. 27 hours in total) over a period of 3 months and one follow up meeting (3 hours) three months after end of treatment. The parents and other relevant close relatives (e.g. siblings, boy/girlfriends) to the patient participate in a workshop where ACT principles are applied. One individual consultation with the adolescent and parents will be offered at the end of 8 sessions of group therapy.
  Arms: Acceptance and Commitment Therapy (ACT)
Other: Enhanced Usual Care (EUC) — All patients will have a thorough clinical psychiatric and somatic assessment in order to determine eligibility and a psychiatric consultation (SPC) of 1-1½ hrs. duration approx. 2 weeks after randomization.
  The consultation is according to a manual and includes psycho-education related to the diagnosis of multiorgan BDS, health promoting recommendations and counselling regarding existing medicine or other treatment. An individualized treatment plan will be sent to the patient's general practitioner, to optimize management in primary care and support by social services.
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
Background:

An increasing number of adolescents report recurrent functional somatic symptoms. Some experience persistent symptoms and may receive functional somatic syndromes (FSS) diagnoses (i.e. symptoms not attributable to any known conventionally defined physical disease), characterised by severe disability and reduced quality of life.

The aim of this study is to:

1. Develop an Acceptance and Commitment Therapy (ACT)-based group intervention for adolescents with severe FSS (conceptualized as Bodily Distress Syndrome (BDS), see detailed description).
2. Examine the efficacy of group based ACT in adolescents (aged 15-19 years) with severe FSS.

The ACT-based treatment, with 9 sessions of group therapy and one follow up meeting is compared to standard treatment/enhanced usual care, which is one single advisory consultation.

The study includes approximately 120 patients.

DETAILED DESCRIPTION:
Background:

An increasing number of adolescents report daily physical symptoms, with a current prevalence of 25%. A substantial proportion of these young people is examined in the health care system, most often with the conclusion that their symptoms cannot be explained in terms of a well-defined medical disease and are hence "stress-related" or "functional". Typically, the symptoms remit spontaneously after the patient is reassured. However, approximately 5-10% experience persistent symptoms and reduced functioning. They may receive diagnoses for functional somatic syndromes (FSS) such as chronic fatigue syndrome (CFS), fibromyalgia (FM), recurrent abdominal pain/irritable bowel syndrome (IBS) or idiopathic pain syndrome. These adolescents are at risk of social isolation, long term school-absence and reduced quality of life.

The aetiology of FSS is assumed complex, with interacting biological, psychological and environmental factors. Recent studies suggest that dysfunction of the stress-axes (e.g. the hypothalamic-pituitary-adrenal (HPA) axis and the autonomic nervous system) and activated inflammatory response are likely to play a role in the development and perpetuation of the symptoms in various FSS. Besides common pathophysiological mechanisms, FSS also show similarities in patient characteristics and treatment response, which speaks in favour of a common family of disorders. Recently, the unifying diagnostic category Bodily Distress Syndrome (BDS) was introduced. BDS is conceptualized as a (patho)physiologic response to prolonged or severe mental and/or physical stress in genetically susceptible individuals, and the diagnosis has been shown to encompass the majority of FSS.

FSS in adults can be managed effectively be means of psychological treatment, but the evidence for adolescents with severe FSS is sparse. Family based cognitive behavioural therapy (CBT) and internet-delivered CBT has proven effective for young patients with particular symptom profiles. However, the development of various specific treatments for each FSS or symptom profile is not an efficient strategy. Recent studies suggest that adult patients with various FSS sampled by the BDS diagnosis can feasibly be treated together, regardless of their main somatic complaint. The same may be true for adolescents, and hence the development of a common treatment for adolescents with various FSS or BDS may be advantageous, and facilitate further implementation in routine clinical care if the treatment is found effective.

Acceptance and Commitment Therapy (ACT), which derives from CBT, has shown promising results in children with chronic functional pain. Improvement could be demonstrated by less avoidance of important activities, better emotional wellbeing and less health care utilization. The aim of this project is to develop an ACT-based group intervention for adolescents with a range of FSS, i.e. conceptualised as severe BDS, and to evaluate its efficacy in a randomized controlled trial.

Method:

Patient population: 120 adolescents with BDS referred to The Research Clinic for Functional Disorders and Psychosomatics (FFL), Aarhus University Hospital. Patients are referred from general practitioners, specialists and hospital wards.

Diagnostic assessment: BDS will be diagnosed after a diagnostic work-up by a physician based on: 1) a review of former medical discharge letters, medical records and other relevant information, 2) SCAN (Schedules for Clinical Assessment in Neuropsychiatry) which screens for general psychopathology and contains a detailed section on BDS 3) screening for ADHD, autism and conduct disorder with screening questions from the child and adolescent psychiatric interview DAWBA (Development and Well Being Assessment), 4) a physical/neurological examination and 5) standard blood tests.

Procedure: Eligible patients, meeting all study criteria, are asked to participate in the RCT. The outcome measures will be filled in at baseline (T0), (i.e. at clinical assessment), before start of therapy (T1), (i.e. two months after baseline), after 8 sessions of therapy (T2), (i.e. 4 months after baseline), two weeks after 9 sessions of therapy (end of treatment, T3) (i.e. 5½ months after baseline) and at eight (T4) and twelve months (T5) after baseline. A physiological assessment of stress response and inflammatory response will be performed at T0 and T5.

Hypotheses:

Primary hypothesis: Patients randomized to ACT-based group therapy will report statistically and clinically significant better self-reported physical health twelve months after baseline, compared to patients receiving a standard psychiatric consultation only (SPC).

Secondary hypotheses: Compared to the control group (SPC), patients receiving ACT-group therapy will at eight and twelve months after baseline: 1. Report statistically and clinically significant reductions in somatic symptoms. 2. Report statistically and clinically significant lower symptom interference and at twelve months after baseline: 3. Show significant improvement in alterations of stress response and inflammatory response. The patients receiving ACT-group therapy will show good feasibility regarding treatment.

ELIGIBILITY:
Inclusion Criteria:

* Severe Bodily Distress Syndrome (multi-organ type) of at least 12 months duration.
* 15-19 year-old.
* Born in Denmark or by Danish parents. Understand, speak and read Danish.

Exclusion Criteria:

* No informed consent.
* An acute psychiatric disorder demanding other treatment, or if the patient is suicidal.
* A lifetime diagnosis of psychosis, mania or depression with psychotic symptoms (ICD-10: F20-29, F30-31, F32.2, F33.3), serious cognitive deficits or developmental disorders such as mental retardation and autism (ICD-10: F70, F84).
* Abuse of narcotics, alcohol or medicine.
* Pregnancy at the time of inclusion.
* Not fit for group based treatment, e.g. patients with severe ADHD (ICD-10: F90), severe social phobia (ICD-10: F40.1) or conduct disorder (ICD-10: F91).

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 91 (Actual)
Dates: Start 2015-01-30 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Change in SF36 (Assessment of physical health) | At baseline (i.e. at clinical assessment) and 2, 4, 5½, 8 and 12 (primary endpoint) months after baseline.
  Questionnaire, patient rated. Physical health measured with aggregate scores of the scales PF (physical functioning), BP (bodily pain) and VT (vitality).

SECONDARY OUTCOMES:
Change in BDS checklist (Assessment of symptom severity) | At baseline (i.e. at clinical assessment) and 12 months after baseline (primary endpoint).
  Questionnaire, patient rated. Assessment of symptom severity.
Change in SCL-somatization Questionnaire (Assessment of functional symptoms) | At baseline (i.e. at clinical assessment) and 2, 4, 5½, 8 and 12 (primary endpoint) months after baseline.
  Questionnaire, patient rated. Assessment of functional symptoms.
Change in Limitation index Questionnaire (Assessment of symptom interference) | At baseline (i.e. at clinical assessment) and 5½, 8 and 12 months after baseline (primary endpoint).
  Questionnaire, patient and parent rated. Assessment of symptom interference.
PGIC (Patient Global Impression of Change) | At 5½, 8 and 12 (primary endpoint) months after baseline.
  Questionnaire, patient and parent rated.
Change in SF36 Questionnaire (Assessment of health related quality of life) | At baseline (i.e. at clinical assessment) and 2, 4, 5½, 8 and 12 (primary endpoint) months after baseline.
  Questionnaire. Patient rated. Assessment of health related quality of life using Social Functioning Scale and Mental Health Scale.
Change in SCL-8, SCL-6, SCL-4 Questionnaire (Assessment of depression and anxiety) | At baseline (i.e. at clinical assessment) and 5½, 8 and 12 (primary endpoint) months after baseline .
  Questionnaire, patient rated. Assessment of depression and anxiety.
Change in HRV heart rate variability (assessment of stress response in various situations (resting state, standing, slow breathing and valsalva) | At baseline (i.e. at clinical assessment) and 12 months after baseline (primary endpoint).
  Physiological assessment of stress response in various situations (resting state, standing, slow breathing and valsalva).
Change in hair cortisol (Measurement of the level of stress-hormone cortisol in hair) | At baseline (i.e. at clinical assessment) and 12 months after baseline (primary endpoint).
  Measurement of the level of stress-hormone cortisol in hair.
Change in level of inflammatory and oxidative stress | At baseline (i.e. at clinical assessment) and 12 months after baseline (primary endpoint).
  Biomarkers for inflammatory and oxidative stress (e.g. IL1, IL6, TNF-alpha, high-sensitive CRP, neopterin, CD163, HO1, MCP1 but also newer proteo-based markers).
Level of physical activity (Anthropometric measurements with accelerometer (Actigraph GT3X) | At baseline (i.e. at clinical assessment) and 12 months after baseline (primary endpoint).
  Anthropometric measurements with accelerometer (Actigraph GT3X), duration 1 week (24h/day).
Change in PSS (Perceived Stress Scale) | At baseline (i.e. at clinical assessment) and 12 months after baseline (primary endpoint).
  Questionnaire, patient rated. Assessment of self perceived stress level.

OTHER OUTCOMES:
Change in AFQ-Y8 (Avoidance and Fusion Questionnaire in Youth) | At baseline (i.e. at clinical assessment) and 2, 4, 5½, 8 and 12 (primary endpoint) months after baseline.
  Questionnaire, patient rated. Assessment of psychological flexibility. Process measure.
Change in IPQ-R Illness Perceptions Questionnaire | At baseline (i.e. at clinical assessment) and 2, 4, 5½, 8 and 12 (primary endpoint) months after baseline.
  Questionnaire, patient rated. Process measure.
Change in BRIQ Behavioural Responses to Illness Questionnaire | At baseline (i.e. at clinical assessment) and 2, 4, 5½, 8 and 12 (primary endpoint) months after baseline.
  Questionnaire, patient rated. Assessment of illness related behaviour. Process measure.
FAD Family Assessment Devise | At baseline (i.e. at clinical assessment) and 12 months after baseline (primary endpoint).
  Questionnaire, patient and parent rated. Assessment of general family functioning. Moderator.
ESQ Experience of Service Questionnaire | 5½ months after baseline (end of treatment).
  Questionnaire, patient rated. Only given to patients in group based therapy. Assessment of their treatment experience.
Change in Whiteley 8 (Assessment of health anxiety) | At baseline (i.e. at clinical assessment) and 2, 4, 5½, 8 and 12 (primary endpoint) months after baseline.
  Questionnaire, patient rated. Assessment of health anxiety. Process measure.
Change in PIPS-12 Psychological Inflexibility in Pain Scale | At baseline (i.e. at clinical assessment) and 2, 4, 5½, 8 and 12 (primary endpoint) months after baseline.
  Questionnaire, patient rated. Assessment of psychological inflexibility. Process measure.
ECR-RS Experience in Close Relationships - relationship structure | At baseline (i.e. at clinical assessment)
  Questionnaire, patient rated. Assessment of attachment style. Moderator.
Credibility/ expectancy questionnaire (Assessment of credibility regarding treatment) | App. two weeks after baseline (i.e. at standard psychiatric consultation (SPC))
  Questionnaire, patient rated. Assessment of credibility regarding treatment.
Life events Questionnaire (Registration of major negative life events) | At baseline (i.e. at clinical assessment)
  Questionnaire, patient rated. Registration of major negative life events.
Other treatment questionnaire (Registration of other received treatment (pharmacological, physiotherapy e.g.) | 12 months after baseline (primary endpoint).
  Questionnaire, patient rated. Registration of other received treatment (pharmacological, physiotherapy e.g.) during the follow-up period.
Registration of adverse events | 12 months after baseline (primary endpoint).
  Questionnaire, patient rated. Registration of potential adverse events during follow up period.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte U Rask, MD, PhD, Principal Investigator — Research Clinic for Functional Disorders and Psychosomatics, Aarhus University Hospital
Locations (1):
- Research Clinic for Functional Disorders and Psychosomatics, Aarhus, Denmark

REFERENCES:
- [Derived] Nyengaard R, Kallesoe KH, Rimvall MK, Ornbol E, Wellnitz KB, Olsen EM, Wyller VBB, Rask CU. Hair cortisol and self-perceived stress in adolescents with multi-system functional somatic disorders. BMC Psychiatry. 2024 Feb 5;24(1):101. doi: 10.1186/s12888-024-05518-4. PMID 38317120
- [Derived] Kallesoe KH, Schroder A, Jensen JS, Wicksell RK, Rask CU. Group-based Acceptance and Commitment Therapy (AHEAD) for adolescents with multiple functional somatic syndromes: A randomised trial. JCPP Adv. 2021 Dec 8;1(4):e12047. doi: 10.1002/jcv2.12047. eCollection 2021 Dec. PMID 37431406
- [Derived] Kallesoe KH, Schroder A, Wicksell RK, Fink P, Ornbol E, Rask CU. Comparing group-based acceptance and commitment therapy (ACT) with enhanced usual care for adolescents with functional somatic syndromes: a study protocol for a randomised trial. BMJ Open. 2016 Sep 15;6(9):e012743. doi: 10.1136/bmjopen-2016-012743. PMID 27633643
- See also: Homepage for the Research Clinic for Functional Disorders, Aarhus University Hospital — http://www.functionaldisorders.dk